CLINICAL TRIAL: NCT04781933
Title: Interest in "Combo" (a Combination of Dietary Supplements Including Probiotics) in NASH Improvement
Acronym: ICAN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mativa-Tech SA (Industry)
Responsible Party: Principal Investigator, Hervé Hagege, Pr, Centre Hospitalier Intercommunal Creteil
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ICAN
Record Dates: First submitted 2021-02-17; First posted 2021-03-04 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: NASH - Nonalcoholic Steatohepatitis
Keywords: Combo; liver stiffness; gut microbiota; dietary supplements
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment with Combo (Active Comparator): 3 dietary supplements will be given
  Interventions: Dietary Supplement: Treatment with Combo
- Treatment with Placebo (Placebo Comparator): 3 placebos will be given
  Interventions: Other: Treatment with placebo

INTERVENTIONS:
Dietary Supplement: Treatment with Combo — Treatment with Combo
  Arms: Treatment with Combo
Other: Treatment with placebo — Treatment with placebo
  Arms: Treatment with Placebo

SUMMARY:
The aim of this bicentre, prospective, placebo-controlled, double-blind, randomized, interventional study is to assess for the first time the effects of a Combo with probiotics and dietary supplements compared to placebo for non-alcoholic steatohepatitis (NASH) patients with mild or severe fibrosis.

DETAILED DESCRIPTION:
Liver-related mortality is increased 10-fold in NASH patients compared with the general population. Currently, there are no established pharmacotherapies for NASH patients. The gut microbiota has a major contributing role in the development of NASH with leaky gut, inflammation, oxidative stress and impaired microbiota. Restoring the microbiota symbiosys could be a new way of resolution of NASH.

The aim of this trial is to evaluate the efficacy of the Combo, association of probiotics (Lactobacillus rhamnosus GG, Bifidobacterium breve BR03, Lactobacillus plantarum) and Glutamine, Quercetin, Vitamin E, Curcumin, Silybin, Pectin by means of histological resolution of NASH without progression of fibrosis, after 26 weeks (6 months), in 60 NASH patients with mild to severe fibrosis.

To confirm a histological diagnosis of NASH and proof efficacy of the Combo, a liver biopsy will be performed prior to screening as well as at the end of supplemental phase

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of moderate to severe NASH :

  * chronic liver disease: biological abnormalities for more than 6 months characteristic ultrasound aspects
  * metabolic syndrome
  * liver stiffness assessed by FibroScan between 8 and 15kPa
* Adults
* Affiliated to a social security
* Women using effective contraception (hormonal or mechanical) for the duration of the srudy

Exclusion Criteria:

* Pregnancy
* Excessive alcohol consumption (>100g/week)
* Cirrhosis (elastometry > 15kPa)
* hepato-cellular carcinoma
* Hepatitis from Corticosteroids, Methotrexate, Amiodarone, Tamoxifen
* Viral hepatitis
* Auto immune hepatitis
* anticoagulant therapy
* antibiotics in the month prior to inclusion
* allergic to soya, aspirin, fish, E110 dye, Maltodextrin
* poorly controlled diabetes (Glycated Hemoglobin >8%)
* inclusion in a drug interventional trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
NASH reduction: the main expected benefit is resolution of NASH, and no worsening of fibrosis | At 6 months
  Evolution of the SAF score and CAP elastometry, a composite histological score taking into account the improvement of Steatosis, histological activity and liver fibrosis

SECONDARY OUTCOMES:
Initial correlation of NASH parameters (FIB4, NAFLD and liver stiffness) and symbiosis parameters (stool analysis by Shallow Shotgun, biological data specific to symbiosis). | At the screening
Follow up of transaminase levels | At 6 months
Reduction of hepatic steatosis measured by CAP elastometry and Hepatic MRI | At 6 months

OTHER OUTCOMES:
Follow up of Biological Scores (FIB4, NAFLD) throughout the study | At 6 months
Follow up of symbiosis throughout the study, analysis of stool of the microbiota and measurement of the biological parameters of the symbiosis; correlation with the evolution of NASH. | At 6 months
Follow up of metabolic syndrome settings throughout the study : weight, waistline, blood pressure, Glycemia, Insulinemia, Gycated Hemoglonin level, Ferritinaemia, Triglyceridemia, HDL Cholesterol, LDL Cholesterol, Apolipoproteine A1, Homa score. | At 6 months

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre Hospitalier Intercommunal Créteil, Créteil
  - Centre Hospitalier Intercommunal de Villeneuve St Georges, Villeneuve-Saint-Georges

IPD SHARING:
Plan to Share IPD: No